CLINICAL TRIAL: NCT02548039
Title: To Study The Influence Of Pharmacogenomics Factors On Pharmacokinetics And Pharmacodynamics Of Clomiphene In Asian Normogonadotrophic Anovulatory Patients.
Brief Title: To Study The Influence Of Genomic Factors On Metabolism And Effects Of Clomiphene In Asian Normogonadotrophic Anovulatory Patients.
Status: Completed | Type: Observational
Sponsor: KK Women's and Children's Hospital (Other Government)
Collaborators: National Cancer Centre, Singapore (Other)
Responsible Party: Sponsor
Other Study IDs: 2014/RM/001
Record Dates: First submitted 2015-09-08; First posted 2015-09-14 (Estimated); Last update posted 2018-08-07 (Actual); Status verified 2018-06

CONDITIONS: Infertility, Female
Keywords: Anovulatory; Clomiphene
MeSH Terms: conditions — Infertility, Female; Anovulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, serum and Genomic DNA.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Asian Normogonadotrophic Anovulatory Women: Asian women with normal gonadotropin levels but do not ovulate.

SUMMARY:
The purpose of this study is to match the genetic component and clinical attributes of anovulatory patients with response to clomiphene treatment.

By improving our understanding on patient-specific clomiphene response will allow optimization of treatment, reduction of side-effects and shorten the time-to-pregnancy.

DETAILED DESCRIPTION:
Anovulation is the commonest cause for infertility, with clomiphene being the standard treatment. Pharmacogenetic causes of variability in the pharmacokinetics and pharmacodynamics of clomiphene is not well characterized in anovulatory Asian women. Although recent findings suggest that the pharmacokinetics and pharmacodynamics of clomiphene may be influenced by several polygenic pathways involving genes regulating its metabolism (CYP3A4, CYP3A5, CYP2B6, CYP2C8, CYP2C19, CYP2D6), thus contributing significantly to the wide variability in dose-response relationships observed in clinical practice. There has not been objective evidence thus far from an unbiased genome-wide perspective. It is likely that polymorphisms at the CYP cluster of genes encoding for their respective cytochrome proteins may not explain all of the variability with regards to clomiphene's dose-response relationship.

The investigators hypothesize that the pharmacokinetics and pharmacodynamics of clomiphene is under strong control by genetic loci and that these genetic variants could also strongly determine the therapeutic outcome in Asian normogonadotrophic anovulatory patients. The contribution by candidate genes mentioned above will also be clarified in a definitive manner by this study.

ELIGIBILITY:
Inclusion Criteria:

* Women of reproductive age with ovulatory dysfunction desiring pregnancy,
* Willing to discontinue any form of herbal or traditional chinese medicines for at least three weeks before starting Clomiphene
* Ability to provide written and informed consent taken from participating patients, and
* Willingness to cooperate with study instructions

Exclusion Criteria:

* Pregnant at the time of recruitment,
* Ovarian cysts more than 5cm,
* Abnormal menorrhagia at the time of study recruitment,
* Abnormal liver function or active liver disease,
* Presence of neoplastic lesions of any type,
* Primary pituitary or ovarian failure (Type I and III World Health Organisation [WHO] Infertility)
* Patients with previous treatment with ovulation inducing agents such as follicle stimulating hormone (FSH) and luteinising hormone releasing hormone-analogues (LHRH-analogues);
* Infertility due to other endocrine abnormalities such as hyperprolactinaemia, hypo/hyperthyroidism, premature ovarian failure, diabetes or male factor
* Allergy to clomiphene.
* Fallopian tubal pathology (hydrosalpinges, previous salpingectomies)
* Patients on any drugs with potential to interact with CYP2D6 such as the selective serotonin receptor uptake inhibitors (ex. Venlafaxine, paroxitene, fluoxetine)

Ages: 21 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Asian Normogonadotrophic Anovulatory Women
Sampling Method: Non-Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2015-01; Primary Completion 2017-03 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Achievement of successful ovulation | Day 20-23 of menses cycle
  Successful ovulation is defined as a mid-luteal phase serum progesterone level of >20 nmol/L.

CONTACTS AND LOCATIONS:
Overall Officials: Jerry Chan, MB BCh BaO (Hons) MA,FRCOG,PhD, Principal Investigator — KK Women's and Children's Hospital
Locations (1):
- KK Women's and Children's Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ghobadi C, Gregory A, Crewe HK, Rostami-Hodjegan A, Lennard MS. CYP2D6 is primarily responsible for the metabolism of clomiphene. Drug Metab Pharmacokinet. 2008;23(2):101-5. doi: 10.2133/dmpk.23.101. PMID 18445989
- [Background] Rostami-Hodjegan A, Lennard MS, Tucker GT, Ledger WL. Monitoring plasma concentrations to individualize treatment with clomiphene citrate. Fertil Steril. 2004 May;81(5):1187-93. doi: 10.1016/j.fertnstert.2003.07.044. PMID 15136073
- [Background] Murdter TE, Kerb R, Turpeinen M, Schroth W, Ganchev B, Bohmer GM, Igel S, Schaeffeler E, Zanger U, Brauch H, Schwab M. Genetic polymorphism of cytochrome P450 2D6 determines oestrogen receptor activity of the major infertility drug clomiphene via its active metabolites. Hum Mol Genet. 2012 Mar 1;21(5):1145-54. doi: 10.1093/hmg/ddr543. Epub 2011 Nov 22. PMID 22108178